CLINICAL TRIAL: NCT02337257
Title: Periodontal and Cardiometabolic Responses to Vitamin D Intervention in African Americans
Brief Title: Periodontal and Cardiometabolic Responses to Vitamin D Intervention in African Americans With Periodontal Disease
Acronym: GumD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Yanbin Dong, Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00001693
Record Dates: First submitted 2014-12-11; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Periodontal Disease; Vitamin D Deficiency
MeSH Terms: conditions — Periodontal Diseases; Vitamin D Deficiency | interventions — Cholecalciferol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cholecalciferol (Active Comparator): Subjects will take 4000 IU per day for 30 days
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): Subjects will take placebo everyday for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — subjects will receive one pill per day which contains 4000 IU/d for 16 weeks
  Other Names: Vitamin D3
  Arms: cholecalciferol
Drug: Placebo — subjects will receive placebo one pill per day for 16 weeks
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Poor vitamin D status is very common in African Americans. Periodontitis (gum disease) are shown to be related to theincreased risk of cardiometabolic diseases. Vitamin D is freely available and cheap supplement that has shown beneficialeffect in the immune system regulation and maintenance of the cardiovascular health. In this study The investigators hypothesize thatvitamin D supplementation for 16 weeks in African Americans with periodontitis will result in clinical improvement in theirgum health as well as their cardiometabolic risk profile

DETAILED DESCRIPTION:
This is a double-blind placebo-controlled randomized clinical trial of vitamin D supplementation.

The eligible subjects will be assigned to a specific group by random assignment in one of the following two groups:

1. Group 1 who will receive placebo.
2. Group 2 who will receive 4,000 IU vitamin D.

Both groups will receive either the placebo pills or vitamin D supplementation everyday for 16 weeks. At visit 1: a fasting morning urine sample will be collected. Height, weight, hip and waist circumferences will be measured. Automatic and manual blood pressures will be measured in sitting position. Approximately 80 ml of venous blood will be collected. Arterial stiffness will be assessed non-invasively by the SphygmoCor device. This device also measures the central (aortic) BP and simultaneously measures pulse wave velocity (PWV). A bottle of 30 capsules containing either vitamin D or placebo will be given to the subjects and will be asked to take one capsule every day for next month till the second visit. A questionnaire to assess the dietary habits, tobacco use, sun exposure, physical activity, socio-economic status and family health history will be given to the subject. At the dental clinic, full mouth clinical measurements (periodontal probing) will be performed. A plaque sample will be taken and a gum biopsy will be taken to examine the dendritic cells. Also, a saliva sample will be collected.

At visit 2: one month later, the supplements will be replenished, compliance will be assessed, and subjects will be examined for any potential side effects.

At visit 3: at 8-week follow up, anthropometric measures, blood samples as well as BP and PWV will be measured and the subject will be assessed for clinical improvement in the periodontitis. All the subjects, irrespective of their group assignment will undergo intensive scaling and root planing (S&RP). The supplements will be replenished, compliance will be assessed, and subjects will be examined for any potential side effects.

Another fasting blood draw, BP measurement and PWV will be performed approximately 24 hours after the S&RP. Also, the investigators will collect saliva sample during this visit.

At visit 4: at 12-week follow up, the procedure in this visit are similar to the visit 2.

At visit 5: at 16-week follow up, a post-test evaluation of vitamin D status, cardiovascular phenotypes and periodontitis will be done at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. You are African American
2. You have generalized chronic moderate to severe gum disease (periodontitis)
3. Your age is between 18-60 years.
4. You are not taking any vitamin, mineral or herbal supplements
5. If you are a female, you are not pregnant

Exclusion Criteria:

* Not meeting any of the above

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Periodontal Disease Activity | Baseline, 8 Weeks, 16 weeks.
  Periodontal disease activity will be measured using standard periodontal disease measures of pocket depth, blood on probing, periodontal inflamed surface area, plaque scores, bone loss, and clinical attachment loss
Change in Cardiometabolic Risk Factors | Baseline, 8 Weeks, 24hrs post-Scaling and Root planing, 16 weeks.
  Cardiometabolic risk factors will be measured by pulse wave velocity, central and peripheral blood pressure and glycated hemoglobin (A1C)

SECONDARY OUTCOMES:
Change in Blood Myeloid Dendritic Cells | Baseline, 8 Weeks, 24hrs post-Scaling and Root planing, 16 weeks.
  Relative gene expression (transcripts) in blood myeloid dendritic cells (mDCs) by polymerase chain reaction (PCR) array, validated by protein, of markers of DC homeostasis and atherogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Yanbin Dong, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States